CLINICAL TRIAL: NCT01437865
Title: Non-invasive Nodal Staging in Breast Cancer With MRI Lymphography Using Gadofosveset; a Pilot-study
Brief Title: Gadofosveset for Axillary Staging in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11-2-016
Record Dates: First submitted 2011-09-12; First posted 2011-09-21 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Breast Neoplasms
Keywords: MRI; lymph node metastases; breast cancer; gadofosveset
MeSH Terms: conditions — Breast Neoplasms; Lymphatic Metastasis | interventions — gadofosveset trisodium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gadofosveset enhanced MRI Axilla (Experimental)
  Interventions: Drug: Gadofosveset contrast agent enhanced MRI Axilla

INTERVENTIONS:
Drug: Gadofosveset contrast agent enhanced MRI Axilla — A MRI of the Axilla will be performed before and after administration of a single IV bolus injection of gadofosveset of an equivalent of 0.03 mmol Gd/kg body weight at an injection speed of 1.5 mL/sec., followed by a saline flush of 25 mL at an injection speed of 1.5 mL/sec.
  Other Names: Gadofosveset (Ablavar/Vasovist) EMEA/H/C/000601

SUMMARY:
The aim of this pilot-study is to examine the accuracy of gadofosveset enhanced MRI compared to current nodal staging methods.

The accuracy of MRL will be determined on the basis of a node-to-node matching of imaged nodes to the definitive histopathology. The pathologic examination of the SNLB or ALND will be regarded as the golden standard for nodal involvement.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with histopathologically confirmed invasive breast cancer about to undergo nodal staging.
2. Tumor must be a T2 according the TNM 6-classification.
3. The ultrasound of the axilla must be suspect for nodal metastases.
4. Willing and able to undergo all study procedures
5. Has personally provided written informed consent.

Exclusion Criteria:

1. Age <18
2. History of prior chemotherapy
3. History of prior radiotherapy of the surrounding areas of the axilla.
4. Pregnancy
5. Contra indications for MRI such as pacemaker, aneurysm clips or severe claustrophobia.
6. Allergy to any of the ingredients of Gadofosveset (Vasovist® /Ablavar®)
7. Being unable to give informed consent in person
8. Acute or chronic severe renal insufficiency (glomerular filtration rate <30 mL/min/1.73m2).
9. Acute renal insufficiency of any severity due to the hepato-renal syndrome or in the perioperative liver transplantation period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-09; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The accuracy (sensitivity, specificity, NPV and PPV) of the MRI in predicting the involvement of metastases | Participants will be followed from the moment of first out-hospital clinic vistit untill final breast surgery, an expected average of 4 weeks.
  The main study parameter will be the accuracy (sensitivity, specificity, NPV and PPV) of the MRI in predicting the involvement of metastases in the investigated lymph nodes. Each node will be scored on MRI as 0= benign, 1=malign. These results will be compared with the histopathological results of the SNLB procedure of ALND procedure on an node by node basis. So the accuray can be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: R. Beets - Tan, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center (MUMC) AZM, Maastricht, Netherlands